CLINICAL TRIAL: NCT02688569
Title: Sleep and Pain Intervention for Chronic Widespread Pain Pilot Study
Acronym: SPIN-CWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Christina McCrae, Professor and Chair, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004488HS
Record Dates: First submitted 2016-01-22; First posted 2016-02-23 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Chronic Widespread Pain; Chronic Insomnia
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT-CWP (Experimental): Participants in this condition will receive Cognitive Behavioral Therapy for Chronic Widespread Pain (CBT-CWP)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Chronic Widespread Pain
- Control (No Intervention): Participants in the Control condition will not receive CBT-CWP. They will however, continue completing the weekly assessments.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Chronic Widespread Pain — CBT-CWP in this study involves 4 sessions of one-hour non-drug behavioral intervention. Session 1 involves education about pain and insomnia and the relationship between the two. Participants will also learn sleep hygiene and stimulus control skills. Session 3 involves teaching participants skills to limit non-sleep time in bed and thus increase sleep efficiency. Participants will also learn the relationship between pain and activity. Session 4 involves teaching participants cognitive restructuring and mindfulness skills to manage maladaptive thoughts related to pain and insomnia. Participants will also review the skills they learned and discuss the maintenance of treatment gains.
  Other Names: CBT-CWP
  Arms: CBT-CWP

SUMMARY:
This randomized controlled clinical trial will examine the effects of Cognitive Behavioral Therapy (CBT-) in patients with comorbid chronic widespread pain (CWP) and insomnia.

Specific Aims:

1. To examine the clinical and health characteristics, including sleep, pain, fatigue, cognitive abilities, and cardiovascular health in patients with comorbid CWP and insomnia.
2. To examine changes in the primary clinical outcomes, including chronic pain, complaints of poor sleep, and fatigue compared to the waitlist control (WLC).
3. To examine changes in the secondary clinical outcomes, including mood, daytime functioning, cognitive functioning, and cardiovascular health compared WLC.
4. To examine the mechanistic variables, including arousal (heart rate variability, HRV), CS (thermal response) and neural plasticity (brain function and structure) - compared to WLC.

DETAILED DESCRIPTION:
This randomized controlled clinical trial will examine the effects of CBT in patients with chronic widespread pain and insomnia. Sample will include 20 patients ([18]-65 years) who satisfy criteria for chronic widespread pain and insomnia. Participants will be randomly assigned to CBT or waitlist control. All participants randomized to the cognitive-behavioral interventions will receive 4 treatment sessions (~50 minutes each). Baseline, posttreatment, [& 3-mo.] follow-up assessments will include measures of sleep, pain, thermal pain response, heart rate variability, brain structure and functions, affect, cognitive functioning, cardiovascular health, and substance use.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Be willing to be randomly assigned to either the treatment condition or the control condition
* Be able to read and understand English
* Have Chronic Widespread Pain (CWP) and Insomnia based on the criteria below:

  o CWP:
* Complaints of pain in upper, lower body, on both sides and the back that lasts for 3+ months.
* Not explained by other illnesses except somatic disorders.

  o Insomnia:
* Insomnia complaints for 6+ months
* Occur despite adequate opportunity and circumstances for sleep
* Consist of 1 or more of the following: difficulty falling asleep, staying asleep, waking up too early, nonrestorative sleep
* Daytime dysfunction (mood, cognitive, social, occupational) due to insomnia
* Baseline diaries indicate >30 minutes of sleep latency or wake after sleep onset combined on 6+ nights.

Exclusion Criteria:

* Be unable to provide informed consent
* Be unwilling to undergo randomization
* Be unable to complete forms and implement treatment due to cognitive impairment (Mini Mental State Examination <26)
* Sleep disorder other than insomnia (i.e., sleep apnea [apnea/hypopnea index, AHI >15]; Periodic Limb Movement Disorder-PLMD [myoclonus arousals per hour >15])
* bipolar or seizure disorder
* other major psychopathology except depression or anxiety (e.g., suicidal ideation/intent, psychotic disorders)
* severe untreated psychiatric comorbidity that renders randomization unethical,
* psychotropic or other medications (e.g., beta-blockers) that alter pain or sleep
* participation in any nonpharmacological treatment (including CBT) for pain, sleep, fatigue, or mood outside the current study,
* internal metal objects or electrical devices
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in self-reported ratings of Pain Sensitivity and Pain Unpleasantness on Daily Diaries | Participants will complete the pain ratings daily for 56 days from Baseline to Post-Treatment , and for 14 days in 3-month Follow-Up (Week 21-22)
  Participants will rate how much pain they experience and how unpleasant the pain is on a scale of 1 to 100 on the daily dairies. Analysis will involve examining the trend of changes in these ratings.
Change in pain severity assessed by the McGill Pain Questionnaire | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
  The McGill Pain Questionnaire will be administered three times - baseline, post-treatment, and follow-up. Analysis will involve examining the trend of change in the scores in McGill Pain Questionnaire.
Change in pain-associated disability assessed by the Pain Disability Questionnaire | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
  The Pain Disability Questionnaire will be administered three times - baseline, post-treatment, and follow-up. Analysis will involve examining the trend of change in the scores in Pain Disability Questionnaire.
Change in Self-Reported Bedtime, Wake time, Sleep Onset Latency, Wake After Sleep Onset, Sleep Quality on the Daily Diaries | Participants will complete the sleep questions daily for 56 days from Baseline to Post-Treatment , and for 14 days in 3-month Follow-Up (Week 21-22)
  Participants will answer the following questions on the daily diaries:
  1. I napped for ____________ minutes yesterday.
  2. I napped ______ times yesterday.
  3. I napped in the ___morning ___afternoon ____evening (check all that apply)
  4. I went to bed last night at ____________ AM/PM.
  5. It took me ____________ minutes to fall asleep.
  6. I woke up ____________ times last night.
  7. I was awake for ____________ minutes in the middle of the night.
  8. My final wake up time was ____________ AM/PM.
  9. I got out of bed at ____________ AM/PM.
  10. I would rate my quality of sleep last night as ____________.
  1. very poor 2. poor 3. fair. 4 good 5. Excellent
Change in Bedtime, Wake time, Sleep Onset Latency, and Wake After Sleep Onset measured by Actigraphy | Daily from the start of the study to post-treatment (week1 to week8), two-week daily reports in 3-mo follow up (week21,week22)
  Actiwatch-L (ACT-L; Mini Mitter, Inc.) will be used to obtain a behavioral measure of sleep outcome. ACT-L is a wristwatch-like device that provides long-term monitoring of ambient light exposure and gross motor activity in human subjects. The Actiware-Sleep software provides behavioral estimates for several sleep variables: (1) sleep onset latency-interval between bedtime and sleep start; (2) total sleep time-sum of all sleep epochs within the sleep period; (3) sleep efficiency percentage- ratio of total sleep time to total time spent in bed × 100; and (4) total wake time-sum of all wake epochs within the sleep period.
Change in Insomnia Severity Index | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
  The Insomnia Severity Index will be administered three times - baseline, post-treatment, and follow-up. Analysis will involve examining the trend of change in the Insomnia Severity Index.

SECONDARY OUTCOMES:
Change in heart rate variability | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in Body Mass Index | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in Cognitive Functioning measured by the NIH toolbox Cognitive Domain | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Day-to-day change in Cognitive Functioning measured by the Cognitive Diary | Participants will complete cognitive diary daily for 56 days from Baseline to Post-Treatment , and for 14 days in 3-month Follow-Up (Week 21-22)
Change in daily substance use | Participants will report daily substance use for 56 days from Baseline to Post-Treatment , and for 14 days in 3-month Follow-Up (Week 21-22)
  Participants will answer these questions:
  Drug Used________________ Prescription Drug? Y/N If yes, used as directed? Y/N Amount taken______________ Time taken________________
Change in Thermal Pain Response | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
  Participants will undergo quantitative sensory testing using a contact thermode applied to the volar surface of the forearm. The protocol that will assess both first pain (primarily A-delta function) and second pain (primarily C-fiber input). All thermal stimuli will be delivered using a computer-controlled Medoc Thermal Sensory Analyzer (TSA-2001, Ramat Yishai, Israel).
  Visual Analog Scale (VAS) ratings of 4 graded intensities (45, 47, 49, 51° C) of 5 second temperature stimuli will be obtained in the following fashion: Stimulus presentation will be timed such that no site is stimulated with less than a 3-minute interval to avoid sensitization of the site. Participants will rate 8 stimuli (2 at each intensity) using a VAS for pain intensity anchored at the right end by "the most intense pain imaginable." A second random sequence of 8 stimuli (2 at each intensity) will be rated by VAS for pain unpleasantness.
Change in food habits measured by 24-hour dietary recall | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in waist-to-hip ratio | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in blood pressure | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in alcohol use frequency as measured by the Alcohol Use Questionnaire | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in alcohol problems as measured by the Alcohol Use Disorders Identification Test | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in grey matter volume as measured by Structural MRI | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in cortical thickness as measured by Structural MRI | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)
Change in functional connectivity in response to thermal pain stimuli as measured by Functional MRI | Pre-treatment (week1 or 2), post-treatment (week7 or 8), follow-up (week 21 or 22)

CONTACTS AND LOCATIONS:
Overall Officials: Christina S McCrae, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- Department of Health Psychology, University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atkinson, J. H., Ancoli-Israel, S., Slater, M., Garfin, S. R., & Gillin, J. C. (1988). Subjective sleep disturbance in chronic pain. Clinical Journal of Pain, 4, 225-232.
- [Background] Currie SR, Wilson KG, Pontefract AJ, deLaplante L. Cognitive-behavioral treatment of insomnia secondary to chronic pain. J Consult Clin Psychol. 2000 Jun;68(3):407-16. doi: 10.1037//0022-006x.68.3.407. PMID 10883557
- [Background] McCrae CS, McGovern R, Lukefahr R, Stripling AM. Research Evaluating Brief Behavioral Sleep Treatments for Rural Elderly (RESTORE): a preliminary examination of effectiveness. Am J Geriatr Psychiatry. 2007 Nov;15(11):979-82. doi: 10.1097/JGP.0b013e31813547e6. PMID 17974868